CLINICAL TRIAL: NCT06000319
Title: Prospective Evaluation of Natural Matrix Protein™ (NMP™) Fibers in Cervical and Lumbar Interbody Fusion
Brief Title: Natural Matrix Protein™ (NMP™) Fibers in Cervical and Lumbar Interbody Fusion
Status: Enrolling by invitation | Type: Observational
Sponsor: Induce Biologics USA Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-NMP-001
Record Dates: First submitted 2023-07-25; First posted 2023-08-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Degenerative Disc Disease; Degenerative Spondylolisthesis; Spinal Stenosis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis | interventions — N-methylpyrrolidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lumbar Interbody Fusion with NMP: Subject has undergone lumbar interbody spine fusion at no more than 3 adjacent levels between L1 and S1 where NMP fibers have been used as a bone void filler
  Interventions: Biological: Natural Matrix Protein (NMP) Fibers; Procedure: Lumbar interbody fusion
- Cervical Interbody Fusion with NMP: Subject has undergone cervical interbody spine fusion at no more than 3 adjacent levels between C2 and T1 where NMP fibers have been used as a bone void filler
  Interventions: Biological: Natural Matrix Protein (NMP) Fibers; Procedure: Cervical interbody fusion

INTERVENTIONS:
Biological: Natural Matrix Protein (NMP) Fibers — human bone allograft
Procedure: Lumbar interbody fusion — Procedure that involves removing the intervertebral disk from the disk space between between 2 or more vertebrae between L1 and S1. When the disk space has been cleared out, the surgeon fills the void between the vertebrae with a bone void filler.
  Groups: Lumbar Interbody Fusion with NMP
Procedure: Cervical interbody fusion — Procedure that involves removing the intervertebral disk from the disk space between between 2 or more vertebrae between C2 and T1. When the disk space has been cleared out, the surgeon fills the void between the vertebrae with a bone void filler.
  Groups: Cervical Interbody Fusion with NMP

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of Natural Matrix Protein™ (NMP™) fibers when used in cervical or lumbar interbody fusion in patients with degenerative disc disease (DDD), spinal stenosis, spondylolisthesis undergoing cervical or lumbar interbody spine fusion at no more than 3 adjacent levels.

DETAILED DESCRIPTION:
The study involves a retrospective review of patients' medical records and prospective collection of X-rays, and patient outcome questionnaires.

The study population will include 100 consecutive lumbar interbody fusion and 100 consecutive cervical interbody fusion patients who meet the inclusion criteria and do not meet the exclusion criteria.

There will be 4 prospective study visits following consent. Follow-up will occur in accordance with standard of care practice and will continue to 12 months post-surgery

ELIGIBILITY:
Inclusion Criteria:

1. Subject was diagnosed with DDD, spinal stenosis, or spondylolisthesis;
2. Subject has undergone cervical or lumbar interbody spine fusion at no more than 3 adjacent levels between C2 and T1 or between L1 and S1;
3. Subject has undergone cervical or lumbar interbody spine fusion using NMP Fibers;
4. Subject must be 18 years of age or older at the time of consent;
5. Subject must be willing and able to sign an informed consent document;
6. Subject must be willing and able to return to the study clinic for all follow-up visits, agree to participate in post-operative clinical and radiographic evaluations.

Exclusion Criteria:

1. Subject is under 18 years of age at the time of consent;
2. Subject is currently experiencing major mental illness (psychosis, schizophrenia, major affective disorder) which in the opinion of the investigator may indicate that the symptoms are psychological rather than of physical origin;
3. Subject is currently imprisoned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include up to 200 patients who have been treated with Induce Biologics NMP™ during cervical or lumbar interbody fusion. All subjects who meet all inclusion criteria and do not meet any exclusion criteria will be included in the study. It is expected that enrollment will take 12 months to complete.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of interbody fusion | Baseline to 12 months post-operative
  Flexion and Extensions radiographs will be assessed for fusion at each level to be fused Fusion is defined as: (1) less than 5 degrees of motion by flexion extension X-ray and (2) no radiological features of non-union (radiolucency, implant migration, loss of graft height, supplemental fixation failure). Both fusion criteria have to be met to be considered a fusion success at the index level.
Incidence of secondary surgical intervention | Baseline to 12 months post-operative
  Secondary surgical interventions (SSI) include revision, re-operation, removal, or supplemental fixation at the index levels
Incidence of Adverse Product Related Events | Baseline to 12 months post-operative
  the incidence of the following will be reported: bone resorption with cage migration or subsidence, local inflammation with seromas, ectopic bone formation, radiculitis.

SECONDARY OUTCOMES:
Incidence of bridging bone | Baseline to 12 months post-operative
  Plane radiographs will be evaluated for the presence of bridging bone at each level to be fused.
Change in disability score for lumbar fusion patients assessed by Oswestry Disability Index | Baseline to 12 months post-operative
  Disability will be assessed using the Oswestry Disability Index (ODI). ODI is a questionnaire to collect a patient's responses to questions about perceived function (disability) in 10 everyday activities in patients with acute or chronic low back pain. Each question consists of 6 statements about 1 activity which are scored from 0 to 5. With 0 indicating the least disability and 5 the greatest. The scores are combined to a single score from 0 (no disability) to 50 (completely disabled)
Change in disability score for cervical fusion patients assessed by Neck Disability Index | Baseline to 12 months post-operative
  Disability will be assessed using the Neck Disability Index (NDI). NDI is a questionnaire to collect a patient's responses to questions about perceived function (disability) in 10 everyday activities in patients with acute or chronic neck pain. Each question consists of 6 statements about 1 activity which are scored from 0 to 5. With 0 indicating the least disability and 5 the greatest. The scores are combined to a single score from 0 (no disability) to 50 (completely disabled)
Change in back pain in lumbar fusion patients | Baseline to 12 months post-operative
  Pain will be assessed by Visual Analogue Scale (VAS) for back pain. VAS is a straight horizontal line of fixed length. The ends are defined as the extreme limits of the pain to be measured from the left (no pain) to the right (worst pain imaginable) and the patient marks on the line how much pain they are experiencing at that time. The VAS score is determined by measuring in millimeters from the end of the line to the point that the patient marks. The minimum score is 0 and the maximum score is 100. The larger the number the worse the pain being experienced
Change in leg pain in lumbar fusion patients | Baseline to 12 months post-operative
  Pain will be assessed by Visual Analogue Scale (VAS) for back pain. VAS is a straight horizontal line of fixed length. The ends are defined as the extreme limits of the pain to be measured from the left (no pain) to the right (worst pain imaginable) and the patient marks on the line how much pain they are experiencing at that time. The VAS score is determined by measuring in millimeters from the end of the line to the point that the patient marks. The minimum score is 0 and the maximum score is 100. The larger the number the worse the pain being experienced.
Change in neck pain in cervical fusion patients | Baseline to 12 months post-operative
  Pain will be assessed by Visual Analogue Scale (VAS) for back pain. VAS is a straight horizontal line of fixed length. The ends are defined as the extreme limits of the pain to be measured from the left (no pain) to the right (worst pain imaginable) and the patient marks on the line how much pain they are experiencing at that time. The VAS score is determined by measuring in millimeters from the end of the line to the point that the patient marks. The minimum score is 0 and the maximum score is 100. The larger the number the worse the pain being experienced.
Change in arm pain in cervical fusion patients | Baseline to 12 months post-operative
  Pain will be assessed by Visual Analogue Scale (VAS) for back pain. VAS is a straight horizontal line of fixed length. The ends are defined as the extreme limits of the pain to be measured from the left (no pain) to the right (worst pain imaginable) and the patient marks on the line how much pain they are experiencing at that time. The VAS score is determined by measuring in millimeters from the end of the line to the point that the patient marks. The minimum score is 0 and the maximum score is 100. The larger the number the worse the pain being experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Prevost Sr, MD, Principal Investigator — Alabama Back Institute; Mark A Prevost II, MD, Principal Investigator — Alabama Back Institute
Locations (1):
- Alabama Back Institute, Jasper, Alabama, United States

IPD SHARING:
Plan to Share IPD: No